CLINICAL TRIAL: NCT03062852
Title: Prévention Des Erreurs médicamenteuses liées Aux Interruptions de tâches Des Soignants Lors de la préparation et de l'Administration Des médicaments : Essai contrôlé randomisé Multicentrique en Clusters
Brief Title: Preventing Drug Errors Related to Caregiver Interruptions
Acronym: PERMIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NI15027; ID-RCB number (Other: 2016-A00211-50); Ministry of Health, France (Other Grant/Funding Number: PREPS-15-000528)
Record Dates: First submitted 2017-02-20; First posted 2017-02-23 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Medication Administered in Error
Keywords: Medication Errors/prevention & control; Nursing Staff, Hospital/organization & administration; Drug Therapy/nursing; Safety Management; Medication Systems, Hospital/organization & administration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medication safety vest (Experimental): During administration rounds, nurses will wear the medication safety vest.
  Interventions: Device: Medication safety vest
- Control (No Intervention): During administration rounds, nurses will be dressed as usual without a safety vest.

INTERVENTIONS:
Device: Medication safety vest — The nurses preparing and administering medication will wear a medication safety vest. On the back of the vest, the sentance "Do not disturb me. I am preparing medications" is written to inform others professional, patients and visitors. A informational flyer will be put in the units to inform patients and visitors about the intervention.
  Arms: Medication safety vest

SUMMARY:
Serious medication administration errors are common in hospitals and nurse's interruptions during medication preparation and administration is associated with errors. Various interventions were developed to help prevention of errors such as visual intervention. Investigators aimed to study the effect of a medication safety vest to reduce medication errors. The vest serves as a visible signal to inform others that the nurse is preparing and administering medications and should not be disturbed. Patients and visitors are provided with an informational flyer to inform them about the use of medication safety vests.

The hypothesis is that the vest will reduce nurse's interruptions during medication preparation and administration, and ultimately reduce medication errors.

The study is a randomized controlled trial in 30 care units of four hospitals in France. Each unit will be randomized in either the control group or the experimental group using the medication safety vest. Nurses of the unit will be selected at random to determine who will be observed during the administration rounds.The observation method will be used to evaluate the error rates in the 2 groups. The number of interruptions and error rates will be evaluated.

DETAILED DESCRIPTION:
Serious medication administration errors are common in hospitals. Significant association between medication administration errors rate and the frequency of nurse's interruptions was shown. The estimated risk of error without interruption during preparation and administration is 2.3% whereas it doubles with 4 or more interruptions.

Various interventions were developed to help prevention of errors such as visual interventions and technology interventions.

Investigators aimed to study the effect of a medication safety vest to reduce medication errors. The vest serves as a visible signal to inform others that the nurse is preparing and administering medications and should not be disturbed. On the back of the vest is written "Do not disturb me. I am preparing medications". Patients and visitors are provided with an informational flyer to inform them about the use of medication safety vests The hypothesis is that the vest will reduce nurse's interruptions during medication preparation and administration, and ultimately reduce medication errors.

The study is a randomized controlled trial in 30 care units of four hospitals in France. Each unit will be randomized in either the control group or the experimental group using the medication safety vest. Nurses of the unit will be randomized to determine who will be observed during the administration rounds.The observation method will be used to evaluate the error rates in the 2 groups. The number of interruptions and error rates will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

- Voluntary nurses of the 30 care units who have drugs to deliver during medication administration rounds will be included.

Exclusion Criteria:

* Nurses who refuse to be observed during medication administration rounds and nurses replacement that did not work usually in the studied units will not be included.
* Nurses in the European G. Pompidou hospital who work in the 4 units involved in an other research project.
* Medication administrations during emergencies (e.g., cardiopulmonary resuscitation) will also be excluded from this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15000 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-04-17 (Actual); Study Completion 2018-04-17 (Actual)

PRIMARY OUTCOMES:
Medication administration errors rate | two weeks after implementation of the medication safety vests and flyers
  The primary outcome is the medication errors rate measured by the observation technique (technique of reference).
  Observers will follow nurses during drug distribution (preparation and administration) to patients, without knowing the physician's medication orders, and will record details about the drugs and interruptions. After completing the observation session, medication administration errors will be assessed blinded to the unit allocation, by comparing the observed medication administered to the medication intended for that patient. The rate of medication administration errors will be calculated by dividing the number of preparation/administration with at least one error by the total opportunities for errors (TOE).

SECONDARY OUTCOMES:
Percentage of wearing medication safety vest | two weeks after implementation of the medication safety vests and flyers
  Observers will note if the nurse is wearing the medication safety vest when arrival in the unit to observe the drug distribution.
Type of medication errors | two weeks after implementation of the medication safety vests and flyers
  Each administration error will be classified by senior pharmacists according to the type of error using the ASHP classification in 9 categories.
Description of nurse's interruptions | two weeks after implementation of the medication safety vests and flyers
  During the drug distribution, the observers will note if the nurse is interrupted and by who. An interruption is defined as a stop in the nurse's task during the medication process and will be classified in 10 categories using the classification from Relihan.
Percentage of nurse's interruptions | two weeks after implementation of the medication safety vests and flyers
  During the drug distribution, the observers will note if the nurse is interrupted. An interruption is defined as a stop in the nurse's task during the medication process and will be classified in 10 categories using the classification from Relihan.
Severity of error | two weeks after implementation of the medication safety vests and flyers
  Each error will be classified by a multidisciplinary committee according to the potential harm using the australian classification from Westbrook in 5 categories.

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Sabatier, PharmD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris (AP-HP)
Locations (1):
- AP-HP, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berdot S, Sabatier B, Gillaizeau F, Caruba T, Prognon P, Durieux P. Evaluation of drug administration errors in a teaching hospital. BMC Health Serv Res. 2012 Mar 12;12:60. doi: 10.1186/1472-6963-12-60. PMID 22409837
- [Background] Berdot S, Gillaizeau F, Caruba T, Prognon P, Durieux P, Sabatier B. Drug administration errors in hospital inpatients: a systematic review. PLoS One. 2013 Jun 20;8(6):e68856. doi: 10.1371/journal.pone.0068856. Print 2013. PMID 23818992
- [Background] Berdot S, Roudot M, Schramm C, Katsahian S, Durieux P, Sabatier B. Interventions to reduce nurses' medication administration errors in inpatient settings: A systematic review and meta-analysis. Int J Nurs Stud. 2016 Jan;53:342-50. doi: 10.1016/j.ijnurstu.2015.08.012. Epub 2015 Sep 7. PMID 26365701
- [Background] Westbrook JI, Woods A, Rob MI, Dunsmuir WT, Day RO. Association of interruptions with an increased risk and severity of medication administration errors. Arch Intern Med. 2010 Apr 26;170(8):683-90. doi: 10.1001/archinternmed.2010.65. PMID 20421552
- [Background] Relihan E, O'Brien V, O'Hara S, Silke B. The impact of a set of interventions to reduce interruptions and distractions to nurses during medication administration. Qual Saf Health Care. 2010 Oct;19(5):e52. doi: 10.1136/qshc.2009.036871. Epub 2010 May 28. PMID 20511596
- [Derived] Berdot S, Vilfaillot A, Bezie Y, Perrin G, Berge M, Corny J, Thi TTP, Depoisson M, Guihaire C, Valin N, Decelle C, Karras A, Durieux P, Le LMM, Sabatier B. Effectiveness of a 'do not interrupt' vest intervention to reduce medication errors during medication administration: a multicenter cluster randomized controlled trial. BMC Nurs. 2021 Aug 24;20(1):153. doi: 10.1186/s12912-021-00671-7. PMID 34429095